CLINICAL TRIAL: NCT00490763
Title: Active Surveillance in Prostate Cancer: A Prospective Cohort Study
Brief Title: Active Surveillance in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2005-0619; R21CA223527-01 (NIH)
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; Prostate Specific Antigen; Questionnaire; Survey
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active Surveillance: Patients with low-risk prostate cancer who choose to undergo active surveillance.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — 7 surveys at the beginning of the study and again every 6 months about diet, coping with the disease, and quality of life.
  Other Names: Questionnaire

SUMMARY:
The goal of this clinical research study is to find out if men who have a type of prostate cancer that has been classified as "low risk" can safely not be treated for the disease. Doctors want to know if patients with "low risk" cancer can avoid or postpone therapy and the related side effects and still live as long as patients who immediately receive therapy.

This is an investigational study. There are no medications used in this trial.

About 1,000 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
You have an early stage of prostate cancer that can be treated effectively with surgery or radiation. If you choose to take part in this study, you will be agreeing to receive only active surveillance. Active surveillance is an investigational way to manage low-stage small volume prostate cancer. While on active surveillance, you will have no treatment for the prostate cancer. However, you will have repeated Prostate Specific Antigen (PSA) tests, physical exams, and other testing to detect when the cancer is becoming a greater risk which may require you to begin treatment.

If you agree to participate in this study, you will not have standard therapy for prostate cancer. Your diagnosis will be confirmed as being of low risk by tests at MD Anderson. Blood will be drawn for PSA tests at the beginning of the study and every 6 months to monitor your cancer.

You will have a biopsy of the prostate at the beginning of the study. Additional prostate biopsies will be performed at your first repeat biopsy at Year 1, and when a doctor thinks it is necessary.

You will have digital rectal examination every 6 months to see if your doctor can feel any prostate nodules. You will have a transrectal ultrasonography every 12 months to see if your doctor can detect any abnormalities in the prostate.

Additionally, you will fill out 7 surveys at the beginning of the study and again every 6 months about how you are coping with the disease and the quality of your life. Each survey will take 5 to 10 minutes to complete.

While you are on study, if an exam or test results show that your disease is getting worse, you will be given the opportunity to have treatment to remove the cancer. If you do choose to receive treatment, you will be taken off study and continue to receive standard follow-up.

Long-Term Follow-Up:

Every 12 months, the study staff will review your medical record or you will be called or e-mailed and asked how you are doing. If you are called, the call would only last a few minutes.

This is an investigational study. About 1,000 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have histologic proof of adenocarcinoma of the prostate within six months of study entry.
2. Patients must agree to have repeat extended 11-core multisite biopsy (sextant locations, midline, and 2 cores each from the left and right anterior horn) of the prostate at study entry. A baseline prostate biopsy is not indicated if a repeat biopsy following the extended biopsy scheme (at least 10 biopsy cores) was performed at The University of Texas M. D. Anderson Cancer Center (MDACC) within 6 months of study entry.
3. Patients who have clinically localized cancer defined by pathologic and PSA criteria to be very low-risk/low-risk, patients with clinically localized cancer [not low-risk] who have refused early intervention or chosen active surveillance as a management option, and patients with clinically localized cancer who are precluded from local therapy because of comorbidities.
4. Patients must agree to comply with the surveillance schedule.
5. Non-English speaking patients may participate in the study, but they will not be required to complete the surveys.
6. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

1. Active noncutaneous malignancy at any site.
2. Prior radiation therapy for treatment of the primary tumor.
3. Planned concomitant immunotherapy, hormonal therapy, chemotherapy, or radiation therapy while on protocol.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with low-risk prostate cancer who choose to undergo active surveillance.
Sampling Method: Probability Sample
Enrollment: 1139 (Actual)
Dates: Start 2006-02-13 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression of Asymptomatic Patients with Clinically Localized Prostate Cancer | 5 years
  Primary end point of the study is time to disease progression, where progression is defined by pathologic criteria and/or an increase in tPSA value.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org